CLINICAL TRIAL: NCT03893539
Title: PRECIsE: A Prospective Evaluation of the Clinical Utility for the Ion Endoluminal System
Brief Title: Clinical Utility for Ion Endoluminal System
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Intuitive Surgical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ISI-ION-001-2018
Record Dates: First submitted 2019-03-26; First posted 2019-03-28 (Actual); Last update posted 2024-03-29 (Actual); Status verified 2024-03

CONDITIONS: Pulmonary Nodule; Lung Cancer; Lung Diseases
MeSH Terms: conditions — Lung Neoplasms; Lung Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Robotic Bronchoscopy (Other): The Ion™ Endoluminal System assists the user in navigating a catheter and endoscopic tools in the pulmonary tract using endoscopic visualization of the tracheobronchial tree for diagnostic and therapeutic procedures. The Ion™ Endoluminal System enables fiducial marker placement. It does not make a diagnosis and is not for pediatric use.
  Interventions: Device: Ion Endoluminal System™

INTERVENTIONS:
Device: Ion Endoluminal System™ — The Ion™ Endoluminal System, Model IF1000, is a software-controlled, electro-mechanical system designed to assist qualified physicians to navigate a catheter and endoscopic tools in the pulmonary tract using endoscopic visualization of the tracheobronchial tree for diagnostic and therapeutic procedures.

SUMMARY:
The goal of this prospective, multi-center, single-arm, clinical study is to evaluate the clinical utility and performance of the FDA-cleared Ion™ Endoluminal System ("Ion") for bronchoscopically approaching and facilitating the tissue sampling of pulmonary nodules.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years and older
* Patient is suitable for elective bronchoscopy
* Patients with a moderate to high risk of lung cancer based on clinical, demographic and radiologic information or with suspected metastatic disease
* Solid or semi-solid pulmonary nodules of ≥ 1cm and ≤ 3cm in largest dimension
* Nodule is located in bronchial generation 4+ (i.e. beyond segmental bronchus*
* Patients are candidates for CT-guided needle biopsy and/or surgical resection
* Patient able to understand and adhere to study requirements
* Patient able to understand and adhere to study requirements and able to provide informed consent
* Patient not legally incapacitated or in legal/court ordered institution
* Patients with no dependency on the investigator or sponsor

Exclusion Criteria:

* Lack of fitness or exercise capacity to undergo bronchoscopy under general anesthesia as determined by physician prior to procedure
* Acute myocardial infarction or unstable angina ≤ 6 weeks prior to study procedure
* Clinically relevant partial trachea obstruction or obstruction of vena cava per physician assessment
* Acute respiratory failure, clinically significant hypoxemia, or high respiratory rate (i.e.> 30 breaths per minute) per physician assessment)
* Renal insufficiency that presents risk per physician's discretion or liver failure (i.e. CHILD-PUGH Class C)
* World Health Organization functional Class III or Class IV Pulmonary Hypertension or history of clinically significant mPAP
* Lung abscess
* Known or suspected pregnancy
* Recent head injury (<12 weeks pre-procedure) or subjects presenting with clinically significant neurologic deficits
* Unstable hemodynamic status (i.e. Dysrhythmia requiring intervention, altered mental status/consciousness)
* Subjects with pure ground glass opacity target nodule
* Inability to adequately oxygenate subject during procedure per physicians discretion (i.e. unable to achieve S02 > 92% or requiring >4L of oxygen prior to procedure)
* Subject with uncorrectable coagulopathy, bleeding or platelet disorders, history of major bleeding with bronchoscopy
* Subjects contraindicated for intubation or general anesthesia, or subjects with ASA ≥ 4
* Subjects taking antiplatelet (i.e. clopidogrel), anti-coagulant (i.e heparin or warfarin) or platelet aggression inhibitors (i.e. Abciximab or Eptifibatide) medications that cannot be stopped per standard practice, i.e. 5-7 days pre-procedure or heparin that cannot be held according to standard practice (6-12 hours). Aspirin not included.
* Any severe or life-threatening comorbidity that could increase the risk of bronchoscopic biopsy (i.e. >Stage 3 heart failure)
* Moderate-to-severe pulmonary fibrosis presenting procedural risk as assessed by physician
* Endobronchial lesion associated with lobar atelectasis
* Presence of bullae >1cm located within a cone based trajectory of biopsy instruments or in location presenting risk per physician assessment
* Known allergy, sensitivity or previous allergic reaction to ortho-phthalaldehyde (OPA)
* Subjects taking the following medications: Immunosuppressive treatment with systemic azathioprine, Cyclosporine, antibodies or cytostatics, other chemotherapeutic agents or medications acting on immunophilins
* Non-systemic treatment for lung cancer (i.e. SBRT, ablation) performed in the same lobe as the target nodule(s)
* Previous surgical intervention (i.e. wedge resection or lobectomy) within the same lobe as target nodule (s)
* Participation in any interventional clinical study or clinical study with experimental agents or agents of unknown risk in last 30 days prior to screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 365 (Actual)
Dates: Start 2019-03-29 (Actual); Primary Completion 2022-05-26 (Actual); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
Navigation Success | Day 1 (Time of Procedure)
Biopsy Success | Day 1 (Time of Procedure)
Sensitivity for Malignancy of System-Obtained Sample | 14 months Post-Procedure

SECONDARY OUTCOMES:
Complications | Intra-procedure, Immediately Post-Procedure, Day 10 Post-Procedure, Day 30 Post-Procedure

CONTACTS AND LOCATIONS:
Overall Officials: Erik Folch, MD, Study Chair — Massachusetts General Hospital
Locations (6):
- United States (6):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconness Medical Center, Boston, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - FirstHealth Moore Regional Hospital, Pinehurst, North Carolina
  - MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Simoff MJ, Pritchett MA, Reisenauer JS, Ost DE, Majid A, Keyes C, Casal RF, Parikh MS, Diaz-Mendoza J, Fernandez-Bussy S, Folch EE. Shape-sensing robotic-assisted bronchoscopy for pulmonary nodules: initial multicenter experience using the Ion Endoluminal System. BMC Pulm Med. 2021 Oct 16;21(1):322. doi: 10.1186/s12890-021-01693-2. PMID 34656103
- [Derived] Agrawal A. Interventional Pulmonology: Diagnostic and Therapeutic Advances in Bronchoscopy. Am J Ther. 2021 Feb 9;28(2):e204-e216. doi: 10.1097/MJT.0000000000001344. PMID 33590989